CLINICAL TRIAL: NCT00752960
Title: DNA Diagnostics for Minimizing Metabolic Side-Effects of Antipsychotics
Acronym: DIMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genomas, Inc (Industry)
Collaborators: Hartford Hospital (Other); University of Kentucky (Other)
Responsible Party: Gualberto Rauno, MD, PhD/President, Genomas, Inc.
Other Study IDs: R44MH073291 (NIH); 50R44 MH073291-03
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Psychoses
Keywords: single nucleotide polymorphism, SNP, aripiprazole, olanzapine, quetiapine, risperidone, ziprasidone, metabolic syndrome
MeSH Terms: conditions — Psychotic Disorders; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- A: Patients receiving olanzapine
- B: patients receiving risperidone
- C: Patients receiving quetiapine
- D: Patients receiving aripiprazole
- E: patients receiving ziprasidone

SUMMARY:
The purpose of this study is to assess patients treated with the antipsychotics aripiprazole (Abilify®), olanzapine (Zyprexa®), quetiapine (Seroquel®), risperidone (Risperdal®), or ziprasidone (Geodon®) and to identify genetic variations more commonly found in individuals who develop diabetic metabolic signs and symptoms, which include changes in blood lipids, blood glucose, blood pressure, and body weight.

DETAILED DESCRIPTION:
As many as 30% of psychiatric patients experience weight gain, central deposition of fat, dyslipidemia, increased blood glucose and hypertension--diabetic metabolic symptoms--upon treatment with atypical antipsychotic medication. As a result, cardiovascular disease risk is significantly increased.

The long-term goal of this collaborative study is to identify, for each individual atypical antipsychotic (AAP) medication, the gene variations associated with elevated risk of diabetic metabolic symptoms (DiMS). If such genes are identified, in the future genetic testing may help mental health care professionals choose treatment while minimizing the risk of undesirable side effects of antipsychotics. We propose to develop a novel product termed "Physiotype" to deliver personalized information for each patient on the drug specific risks among aripiprazole, olanzapine, quetiapine, risperidone, and ziprasidone. The Physiotype consists of a multi-gene ensemble of single nucleotide polymorphisms (SNPs) that, interpreted with a biomathematical algorithm, may explain most of the inter-individual differences in DiMS among the 5 AAPs. If this study does identify related genes, genetic tests will be developed to provide patients and health care professionals with tools to identify those patients who are at risk of developing adverse metabolic side effects to antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* receiving atypical antipsychotic therapy (olanzapine, aripiprazole, quetiapine, risperidone, or ziprasidone) for 3 months
* who have taken >50% of the prescribed dose for the last month.

Exclusion Criteria:

* none

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients treated for psychoses
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
diabetic metabolic symptoms (DiMS): body weight, body mass index, waist circumference, blood pressure, triglycerides, total, LDL, and HDL cholesterol, blood glucose | after treatment with antipsychotic medication(s) for => 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto Ruano, MD, PhD, Principal Investigator — Genomas, Inc
Locations (2):
- United States (2):
  - Hartford Hospital Institute of Living, Hartford, Connecticut
  - University of Kentucky, Lexington, Kentucky

REFERENCES:
- [Background] Ruano G, Blair CL, Bower B, Windemuth A, Kocherla M, Aleman Y, Pearlson G, Goethe JW, Schwartz HI. Somatic complications of psychotropic medications in a patient with multiple CYP2 drug metabolism deficiencies. Conn Med. 2007 Apr;71(4):197-200. PMID 17487003
- [Background] de Leon J, Susce MT, Johnson M, Hardin M, Pointer L, Ruano G, Windemuth A, Diaz FJ. A clinical study of the association of antipsychotics with hyperlipidemia. Schizophr Res. 2007 May;92(1-3):95-102. doi: 10.1016/j.schres.2007.01.015. Epub 2007 Mar 8. PMID 17346932
- [Background] Ruano G, Goethe JW, Caley C, Woolley S, Holford TR, Kocherla M, Windemuth A, de Leon J. Physiogenomic comparison of weight profiles of olanzapine- and risperidone-treated patients. Mol Psychiatry. 2007 May;12(5):474-82. doi: 10.1038/sj.mp.4001944. Epub 2007 Jan 2. PMID 17199131
- [Derived] Windemuth A, de Leon J, Goethe JW, Schwartz HI, Woolley S, Susce M, Kocherla M, Bogaard K, Holford TR, Seip RL, Ruano G. Validation of candidate genes associated with cardiovascular risk factors in psychiatric patients. Prog Neuropsychopharmacol Biol Psychiatry. 2012 Mar 30;36(2):213-9. doi: 10.1016/j.pnpbp.2011.08.001. Epub 2011 Aug 6. PMID 21851846
- See also: Institute of Living, Hartford Hospital, Hartford, CT — http://www.instituteofliving.org/